CLINICAL TRIAL: NCT01127763
Title: Phase II Trial of RAD001 Plus Carboplatin in Patients With Triple-Negative Metastatic Breast Cancer
Brief Title: RAD001 Plus Carboplatin in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU 09-0060
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
Keywords: metastatic; breast; cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Everolimus; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001+carboplatin (Experimental): Carboplatin (starting dose was initially AUC 6, later decreased to AUC 5, then AUC 4) every 3 weeks as IV infusion and RAD001 as 5 mg pill each day until disease progression or unacceptable toxicity.
  Interventions: Drug: RAD001; Drug: Carboplatin

INTERVENTIONS:
Drug: RAD001
  Other Names: Afinitor; Everolimus
Drug: Carboplatin
  Other Names: Paraplatin

SUMMARY:
This study investigates the effectiveness of combination of carboplatin and investigational agent RAD001 in triple-negative breast cancer.

DETAILED DESCRIPTION:
The primary objective of this study was to determine clinical benefit rate (CBR) i.e.complete remission (CR) + partial remission (PR) + stable disease (SD) lasting ≥ 6 months, and the toxicity of RAD001 /carboplatin in women with metastatic triple-negative breast cancer. Treatment consisted of intravenous carboplatin at area under the plasma concentration-time curve (AUC) 6, later decreased to AUC 5, and subsequently to AUC 4 every 3 weeks with daily 5mg RAD001.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer (measurable or evaluable including bone metastases only)
* Histologically confirmed triple negative breast cancer (estrogen receptor (ER)< 10%, progesterone receptor (PR) < 10 %, Her2neu IHC 0 or 1 or FISH negative)
* Age >= 18 years
* World Health Organization performance status <= 2
* Adequate bone marrow function as shown by: absolute neutrophil count ≥ 1.5 x 10^9/L, Platelets ≥ 100 x 10^9/L, Hb >9 g/dL
* Adequate liver function as shown by:

  1. serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  2. international normalized ratio (INR): Patients not on warfarin INR ≤1.5; Patients on warfarin INR ≤3; Patient on stable dose of low molecular weight heparin for >2 weeks at time of treatment is allowed.
  3. alanine aminotransferase and aspartate aminotransferase ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Signed informed consent
* Patients may have had 0-3 prior regimens for metastatic disease and prior bevacizumab (avastin) is allowed.
* A baseline lung CT (or PET/CT)
* O2 sat >= 90% in room air (if <90%, spirometry and diffusion capacity of lung for carbon monoxide (DLCO) above 50% of the normal predicted value of pulmonary function tests)
* Negative serum pregnancy test within 7 days prior to starting treatment

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 2 weeks of the start of study drug (including chemotherapy, radiation therapy, and biologics)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 2 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent, except corticosteroids with a daily dosage equivalent to prednisone ≤ 20 mg. However, patients receiving corticosteroids must have been on a stable dosage regimen for a minimum of 4 weeks prior to the first treatment with RAD001. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  1. Symptomatic congestive heart failure of New York heart Association Class III or IV
  2. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  3. severely impaired lung function as defined as spirometry and DLCO that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  4. uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
  5. active (acute or chronic) or uncontrolled severe infections
  6. liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis. Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA polymerase chain reaction testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Ongoing alcohol or drug addiction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Clinical Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Singh J, Novik Y, Stein S, Volm M, Meyers M, Smith J, Omene C, Speyer J, Schneider R, Jhaveri K, Formenti S, Kyriakou V, Joseph B, Goldberg JD, Li X, Adams S, Tiersten A. Phase 2 trial of everolimus and carboplatin combination in patients with triple negative metastatic breast cancer. Breast Cancer Res. 2014 Mar 31;16(2):R32. doi: 10.1186/bcr3634. PMID 24684785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2010 to July 2012, 25 patients were enrolled from New York University Medical center and its affiliated hospitals.
Period: Overall Study
Arm/Group | RAD001+Carboplatin
Started | 25
Completed | 20 (Patients off study due to disease progression were considered to have completed the study.)
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | RAD001+Carboplatin
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Number of prior chemotherapy regimens [Median (Full Range); unit: chemotherapy regimens] | 1 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (Complete Response, Partial Response, and Stable Disease That Lasts More Than 6 Months)
Description: Clinical benefit rate is defined as the number of patients with complete response (CR), partial response (PR), or stable disease (SD) that lasts at least 6 months. Response was assessed every 2 cycles of treatment (6 weeks) by computed tomography (CT), CT/positron emission tomography (PET), or magnetic resonance imaging (MRI). Overall response evaluation is based on Response Evaluation Criteria In Solid Tumors 1.0 (RECIST 1.0). Per RECIST 1.0 for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: up to 1 year
Population: Any patient with at least one dose of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- RAD001+Carboplatin: Carboplatin (starting dose was initially AUC 6, later decreased to AUC 5, then AUC 4) every 3 weeks as IV infusion and RAD001 as 5 mg pill each day until disease progression or unacceptable toxicity.
  RAD001
  Carboplatin
Arm/Group | RAD001+Carboplatin
Number analyzed (Participants) | 25
percentage of patients | 36 [21 to 57]

2. Primary Outcome: Toxicity Profile-Hematological
Description: Reported as percentage of patients who experienced grade 3 and higher hematological adverse events (AEs) related to the study drugs.
Time Frame: treatment period (up to 1 year) plus 30 days off treatment
Population: any patient who received at least 1 dose of protocol treatment.
Measure: Number; unit: percentage of patients
Groups:
- RAD001+Carboplatin (AUC 6 and 5): Carboplatin (starting dose of AUC 6 or AUC 5) every 3 weeks as IV infusion and RAD001 as 5 mg pill each day.
- RAD001+Carboplatin (AUC 4): Carboplatin (starting dose of AUC 4) every 3 weeks as IV infusion and RAD001 as 5 mg pill each day.
- RAD001+Carboplatin (All Patients): Carboplatin every 3 weeks as IV infusion and RAD001 as 5 mg pill each day.
Arm/Group | RAD001+Carboplatin (AUC 6 and 5) | RAD001+Carboplatin (AUC 4) | RAD001+Carboplatin (All Patients)
Number analyzed (Participants) | 7 | 18 | 25
percentage of patients
  Anemia | 0 | 5 | 4
  Thrombocytopenia | 71 | 11 | 28
  Leukopenia | 14 | 0 | 4
  Neutropenia | 29 | 5 | 12

3. Secondary Outcome: Median Progression-free Survival Time
Description: Progression-free survival time is defined as the time from first day of treatment to the first date of disease progression or death as a result of any cause. Progression was assessed every 2 cycles of treatment (6 weeks) by CT, CT/PET, or MRI. Progression is defined using RECIST 1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 1 year
Population: Any patient with at least one dose of treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001+Carboplatin
Number analyzed (Participants) | 25
months | 3 [2 to 5]

4. Primary Outcome: Toxicity Profile-Non Hematological
Description: Reported as percentage of patients who experienced grade 3 and higher non-hematological AEs related to the study drugs.
Time Frame: treatment period (up to 1 year) plus 30 days off treatment
Population: any patient who received at least 1 dose of protocol treatment.
Measure: Number; unit: percentage of patients
Arm/Group | RAD001+Carboplatin (All Patients)
Number analyzed (Participants) | 25
percentage of patients
  Nausea | 4
  Vomiting | 4
  Dehydration | 4
  Mucositis | 4
  Hypersensitivity | 4

ADVERSE EVENTS:
Time Frame: AEs were assessed during the treatment and 30 days from the last day of treatment.
Description: All AEs are reported here regardless of attribution.
Arm/Group | RAD001+Carboplatin
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001+Carboplatin (N=25)
Hypertension (Cardiac disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils (Infections and infestations) | 2
Pain (Nervous system disorders) | 1
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001+Carboplatin (N=25)
Allergic Reaction/Hypersensitivity (Including Drug Fever) (Immune system disorders) | 1
Hemolysis (E.G., Immune Hemolytic Anemia, Drug-Related Hemolysis) (Blood and lymphatic system disorders) | 9
Leukocytes (Total Wbc) (Investigations) | 4
Neutrophils/Granulocytes (Anc/Agc) (Investigations) | 11
Platelets (Investigations) | 16
Inr (International Normalized Ratio Of Prothrombin Time) (Investigations) | 1
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 11
Fever (In The Absence Of Neutropenia, Where Neutropenia Is Defined As Anc <1.0 X 10e9/L) (General disorders) | 3
Insomnia (Psychiatric disorders) | 1
Bruising (In Absence Of Grade 3 Or 4 Thrombocytopenia) (Injury, poisoning and procedural complications) | 1
Dermatology/Skin - Other (Specify, skin nodules (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4
Rash: Acne/Acneiform (Skin and subcutaneous tissue disorders) | 4
Hot Flashes/Flushes (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 2
Dry Mouth/Salivary Gland (Xerostomia) (Gastrointestinal disorders) | 1
Mucositis/Stomatitis (Functional/Symptomatic) (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Taste Alteration (Dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Hemorrhage, Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 3
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils (Infections and infestations) | 2
Dermal Change Lymphedema, Phlebolymphedema (Blood and lymphatic system disorders) | 2
Edema: Head And Neck (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 4
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3
Alt, Sgpt (Serum Glutamic Pyruvic Transaminase) (Metabolism and nutrition disorders) | 3
Ast, Sgot(Serum Glutamic Oxaloacetic Transaminase) (Metabolism and nutrition disorders) | 2
Cholesterol, Serum-High (Hypercholestremia) (Investigations) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Extremity-Lower (Gait/Walking) (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness, Generalized Or Specific Area (Not Due To Neuropathy) (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 4
Mood Alteration (Nervous system disorders) | 1
Neuropathy: Sensory (Nervous system disorders) | 3
Dry Eye Syndrome (Eye disorders) | 1
Pain - Other (Specify, incisional pain) (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Cavity/Paranasal Sinus Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Voice Changes/Dysarthria (E.G., Hoarseness, Loss Or Alteration In Voice, Laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Vaginal Discharge (Non-Infectious) (Reproductive system and breast disorders) | 1
Pain_extremity-limb (Musculoskeletal and connective tissue disorders) | 3
Pain_joint (Musculoskeletal and connective tissue disorders) | 1
Pain_back (Musculoskeletal and connective tissue disorders) | 4
Pain_headache (Nervous system disorders) | 4
Pain_breast (Reproductive system and breast disorders) | 2
Pain_stomach (Gastrointestinal disorders) | 1
Pain_bone (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No